CLINICAL TRIAL: NCT00621608
Title: A Prospective, Double-blind, Randomized, Controlled Clinical Trial Comparing Standard Wound Care With Adjunctive Hyperbaric Oxygen Therapy (HBOT) to Standard Wound Care Only for the Treatment of Chronic, Non-healing Ulcers of the Lower Limb in Patients With Diabetes Mellitus.
Brief Title: Hyperbaric Oxygen Therapy (HBOT) for Chronic Diabetic Lower Limb Ulcers
Acronym: HBOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Judy Dan Research and Treatment Centre Ontario Wound Care Inc (Unknown); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Ron Goeree, Director, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HTA011-0708-01
Record Dates: First submitted 2008-01-29; First posted 2008-02-22 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus; Chronic Ulcers of the Lower Limb
Keywords: Chronic ulcers; Diabetes; Hyperbaric Oxygen Therapy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Hyperbaric Oxygen Therapy
  Interventions: Procedure: Hyperbaric Oxygen Therapy
- 2 (Sham Comparator): Placebo Hyperbaric Oxygen Chamber
  Interventions: Procedure: Placebo Hyperbaric Oxygen Chamber

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — Hyperbaric Oxygen Therapy (HBOT) will be provided 5 days per week for 6 weeks for a total of 30 treatments on average. Subjects will be placed into the hyperbaric chamber for approximately 90 minutes of HBOT at 2.4 ATA (partial pressure of oxygen = 1,800 mmHg) when inside the chamber. Subjects will receive dressing changes as required per standard of care.
  Arms: 1
Procedure: Placebo Hyperbaric Oxygen Chamber — Patients will receive HBOT placebo 5 days per week for 6 weeks for a total of 30 treatments. Each patient will be placed into the hyperbaric chamber and will receive 90 minutes of room air while inside the chamber and the initial flow of air into the chamber will produce a small increase in pressure (0.3 ATA partial pressure of oxygen = 210 mmHg) which will then be released over a period of 10 minutes. Subjects will receive dressings changes as required per standard of care.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if HBOT plus standard wound care is more effective than standard wound care alone at preventing the need for major amputation (metatarsal and up) in patients with diabetes mellitus (Type 1 or 2) with moderate to sever chronic wounds of lower limbs.

DETAILED DESCRIPTION:
People with diabetes mellitus and non-healing ulcers of the lower limb are at higher risk of amputation. Current standard care for foot ulcers includes maintaining optimal blood glucose levels, use of debridement, antibacterials, dressings, antibiotics for infection; adequate nutrition; pressure relief and amputation. There has been an increased interest in the use of hyperbaric oxygen therapy (HBOT) as an adjunctive treatment for diabetic ulcers. HBOT is an established technology which currently is an accepted treatment of chronic diabetic ulcers in Ontario and physicians who provide this service are reimbursed under the current Ontario Health Insurance Plan (OHIP). However there are only a few facilities that can provide this service. In addition, results of published HBOT studies are inconsistent. The current study will provide quality efficacy data on the use of HBOT as an adjunctive therapy. As this study has been recommended by the Ontario Health Technology Advisory Committee (OHTAC), the results of the study will be used to make policy decisions regarding the funding and further utilization of HBOT therapy for people with diabetes mellitus with ulcers of the lower limb in the province. If the results are favorable towards HBOT in the treatment of diabetic ulcers, potential expansion and availability of this and other programs maybe be possible. A randomized placebo control trial evaluating HBOT, to the best of our knowledge has not been completed in this area and will provide much needed information to the scientific community.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Type 1 or 2 Diabetes Mellitus
* Wagner grading of foot lesions 3 or 4 on lower limb not healing for 4 weeks.

Exclusion Criteria:

* Impending urgent amputation due to ongoing or exacerbated infection;
* Exposed calcaneus bone with no prospect of weight bearing potential even if defect has been healed;
* Dialysis-dependent renal failure;
* Any of the following medical conditions which preclude safe treatment in a monoplace chamber: clinical depression; severe dementia; claustrophobia; seizure disorder; active asthma; severe chronic obstructive pulmonary disease; previous thoracic surgery; previous spontaneous or trauma induced pneumothorax; history of severe congestive heart failure with left ventricular ejection fraction less than 20%; unstable angina; chronic sinusitis; chronic or acute otitis media or major ear drum trauma; severe kyphoscoliosis; arthritis; or morbid obesity;
* History of chemotherapy with use of Bleomycin;
* Participation in another investigative drug or device trial currently or within the last 30 days;
* Current candidates for vascular surgery, angioplasty or stenting;
* Major large vessel disease;
* Undergone vascular surgery or angioplasty within the last 3 months;
* Women who are currently pregnant or are breast feeding or women of childbearing potential who are not currently taking adequate birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-04; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Freedom from having, or meeting the criteria for, a major amputation (below knee amputation, or metatarsal level) up to 12 weeks after randomization. | up to 12 weeks after randomization

SECONDARY OUTCOMES:
Wound healing: difference in wound measurements (i.e. depth, length, width and extent of surface area); reduction in Wagner Classification Score; proportion of wound closed at 12 weeks of any time interval prior to end point; time to healing (days) | up to 12 weeks after randomization
Effectiveness: maintenance on therapy (discontinuation rates); and secondary prevention interventions (confounding variables that may influence primary outcome such as diabetes control) | up to 12 weeks after Randomziation
Safety: Major morbidity (infection requiring hospitalization, renal failure); wound interventions during study (debridement, surgery); Complications related to HBOT (seizure, pulmonary syndromes, vision disturbance; and all cause mortality | From enrollment up to 1 year after randomization
Healthcare resource utilization: wound dressing materials; healthcare provider visits; inpatient hospital admissions; complex continuing care/rehabilitation; drug therapy; mobility assistive devices | From enrollment to study up to 1 year after randomization
Quality of life: assessed by Standard Form 36 (SF-36) domain scores; EuroQoL 5D (EQ-5D) summary scores and by the Diabetic Foot Ulcer-Short Form (DFS-SF) scores | Baseline, end of treatment, end of follow-up, and EQ5D only at 6 and 12 months
Cost effectiveness of HBOT: calculate the incremental cost per amputation avoided and the incremental cost per quality-adjusted life-year (QALY) gained | From Enrollment to 1 year after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Daria O'Reilly, PhD, Study Chair — Programs for Assessment of Technology in Health Research Institute; Ludwik Fedorko, MD, Principal Investigator — Judy Dan Wound Care Centre/University Health Network; Ron Linden, MD, Principal Investigator — Judy Dan Wound Care Centre/University Health Network
Locations (1):
- Judy Dan Wound Care Centre/University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] O'Reilly D, Linden R, Fedorko L, Tarride JE, Jones WG, Bowen JM, Goeree R. A prospective, double-blind, randomized, controlled clinical trial comparing standard wound care with adjunctive hyperbaric oxygen therapy (HBOT) to standard wound care only for the treatment of chronic, non-healing ulcers of the lower limb in patients with diabetes mellitus: a study protocol. Trials. 2011 Mar 7;12:69. doi: 10.1186/1745-6215-12-69. PMID 21385365
- [Derived] Fedorko L, Bowen JM, Jones W, Oreopoulos G, Goeree R, Hopkins RB, O'Reilly DJ. Hyperbaric Oxygen Therapy Does Not Reduce Indications for Amputation in Patients With Diabetes With Nonhealing Ulcers of the Lower Limb: A Prospective, Double-Blind, Randomized Controlled Clinical Trial. Diabetes Care. 2016 Mar;39(3):392-9. doi: 10.2337/dc15-2001. Epub 2016 Jan 6. PMID 26740639